CLINICAL TRIAL: NCT03824028
Title: Post-Market Clinical Survey of Clareon® IOL With the AutonoMe™ Automated Preloaded Delivery System With Japanese Subjects
Brief Title: Post-Market Clinical Survey of Clareon® IOL AutonoMe™ in Japanese Subjects
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: ILM171-P001
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Cataract
Keywords: Cataract surgery; Intraocular lens; IOL; Clareon; AutonoMe
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clareon IOL AutonoMe: Prior implantation with Clareon intraocular lenses (IOLs) using the Clareon® IOL AutonoMe™ automated preloaded delivery system
  Interventions: Device: Clareon® IOL AutonoMe™ automated preloaded delivery system

INTERVENTIONS:
Device: Clareon® IOL AutonoMe™ automated preloaded delivery system — Disposable injector preloaded with the Clareon IOL for precise IOL insertion during cataract surgery

SUMMARY:
This purpose of this survey study is to collect and describe clinical outcomes for the intraocular lens (IOL) delivery performance of Clareon® IOL AutonoMe™ when used in daily practice.

DETAILED DESCRIPTION:
This study will enroll subjects who underwent prior cataract surgery with phacoemulsification and were implanted with Clareon intraocular lenses (IOLs) using the Clareon® IOL AutonoMe™ automated preloaded delivery system. Subjects will be enrolled post-operatively and followed for one year.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign informed consent.
* Prior diagnosis of age-related cataracts.
* Prior cataract surgery with implantation of Clareon IOL in the capsular bag by AutonoMe™.
* No ophthalmic disease which might affect visual acuity.

Exclusion Criteria:

* None.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled at approximately 20 investigative sites located in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Best-corrected distance visual acuity | Up to Year 1 postoperative
  Visual acuity will be collected under well-lit conditions at a distance of five meters using a decimal visual acuity chart.
Intraocular lens (IOL) delivery performance | Surgery day (retrospective)
  A questionnaire will be used to retrospectively evaluate the usability of AutonoME™. The investigator will respond to 8 questions pertaining to the IOL delivery performance using a 5-point scale where 1 = very good/strongly agree and 5 = very poor/strongly disagree.
Difference between target refraction and postoperative subjective refraction (spherical equivalent) | Up to Year 1 postoperative
  Visual acuity will be collected under well-lit conditions at a distance of five meters using a decimal visual acuity chart. Subjective refraction at best corrected distance vision will be recorded and compared with target refraction determined on day of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Japan, Ltd.
Locations (3):
- Japan (3):
  - Alcon Investigative Site, Yokohama, Kanagawa
  - Alcon Investigative Site, Yokkaichi, Mie-ken
  - Alcon Investigative Site, Hashimoto, Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oshika T, Sasaki N; Clinical Study Group on New Intraocular Lens and Delivery System. One-year multicenter evaluation of a new hydrophobic acrylic intraocular lens with hydroxyethyl methacrylate in an automated preloaded delivery system. J Cataract Refract Surg. 2022 Mar 1;48(3):275-279. doi: 10.1097/j.jcrs.0000000000000746. PMID 34261986